CLINICAL TRIAL: NCT03618329
Title: Effect of Prehabilitation on the Lean Mass Index (IMM) in Patients Operated on for Colon Cancer in ERAS Programm.
Brief Title: Effect of Prehabilitation on the Lean Mass Index (IMM) in ERAS PROGRAMM.
Acronym: PRERAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Antonio Arroyo Sebastian, Prof, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRERAS
Record Dates: First submitted 2018-07-31; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Colo-rectal Cancer; Nutrition Disorders
Keywords: COLON CANCER; ERAS; NUTRITION
MeSH Terms: conditions — Colonic Neoplasms; Nutrition Disorders | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Active Comparator): exercise, nutrition and anxiety reduction in the preoperative period
  Interventions: Other: Prehabilitation
- No Prehabilitation (No Intervention): Not: exercise, nutrition and anxiety reduction in the preoperative period

INTERVENTIONS:
Other: Prehabilitation — exercise, nutrition and anxiety reduction in the preoperative period
  Arms: Prehabilitation

SUMMARY:
The implementation of prehabilitation in patients operated on for colon cancer in a multimodal rehabilitation regimen improves the values of the "lean body mass" or lean mass index, positively influencing the results of clinical, analytical and radiological nutritional values pre- and postoperatively and in morbi-mortality, recovery, average stay and re-entry rates.

ELIGIBILITY:
Inclusion Criteria:

* It is considered that the subject suffers a confirmed diagnosis of colon cancer and is going to undergo surgery on a scheduled basis under a RHMM program.
* The subject is ≥ 18 years of age.
* The subject can perform any of the two proposed treatments.
* Preoperative staging TxNxM0.
* The patient has voluntarily signed and dated an informed consent document (IC), approved by an independent Ethics Committee (CEIC) before participating in the study.

Exclusion Criteria:

* Patients with rectal cancer.
* The study doctor determines that the subject is not eligible to participate.
* The subject can not give informed consent to participate in the study.
* The subject can not perform the pre-habilitation.
* Non-acceptance or impossibility of following rehabilitation protocol multimodal
* The subject was previously scheduled at the time of the inclusion of the nutritional supplement study, whether it is different or the same that would be scheduled at this time
* Subjects who have received previous radiochemotherapy, HIV, gestational stage, psychiatric, with CRF who are undergoing renal replacement techniques, urgent surgery, with intestinal obstructions, with uncontrolled infections, urgent surgery, distant metastasis, ASA IV, advanced liver failure, severe coagulation disorder, severe hyperlipidemia and hyperglycemia or difficult to control.
* Subject has renal or hepatic impairment (GFR <60ml / m or AST / ALT 3 x upper limit of normal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Effect of prehabilitation on the change from lean mass index | preoperative and 1-month postoperative
  Effect of prehabilitation on the lean mass index

REFERENCES:
- [Derived] Triguero-Canovas D, Lopez-Rodriguez-Arias F, Gomez-Martinez M, Sanchez-Guillen L, Peris-Castello F, Alcaide-Quiros MJ, Morillas-Blasco P, Arroyo A, Ramirez JM. Home-based prehabilitation improves physical conditions measured by ergospirometry and 6MWT in colorectal cancer patients: a randomized controlled pilot study. Support Care Cancer. 2023 Nov 6;31(12):673. doi: 10.1007/s00520-023-08140-4. PMID 37930478
- [Derived] Lopez-Rodriguez-Arias F, Sanchez-Guillen L, Aranaz-Ostariz V, Triguero-Canovas D, Lario-Perez S, Barber-Valles X, Lacueva FJ, Ramirez JM, Arroyo A. Effect of home-based prehabilitation in an enhanced recovery after surgery program for patients undergoing colorectal cancer surgery during the COVID-19 pandemic. Support Care Cancer. 2021 Dec;29(12):7785-7791. doi: 10.1007/s00520-021-06343-1. Epub 2021 Jun 24. PMID 34169328